CLINICAL TRIAL: NCT04479163
Title: Prevention of Severe Covid-19 in Infected Elderly by Early Administration of Convalescent Plasma With High-titers of Antibody Against SARS-CoV2.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Infant (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FundacionINFANT-Plasma
Record Dates: First submitted 2020-06-29; First posted 2020-07-21 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: COVID

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma (Experimental): Convalescent plasma with an IgG titer against SARS-CoV2
  Interventions: Biological: Convalescent Plasma
- Placebo (Placebo Comparator): Normal Saline 0.9%
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Convalescent Plasma — 250 ml Convalescent plasma with an IgG titer against SARS CoV2
  Arms: Plasma
Other: Placebo — Normal Saline 0.9%
  Arms: Placebo

SUMMARY:
Trial design. Randomized, double-blind, placebo-controlled trial in a catchment population of 2,020,860 age-appropriate subjects in the state of Buenos Aires and 235,000 in the city of Buenos Aires.

Institutions. Hospitals San Juan de Dios, Simplemente Evita, Dr. Carlos Bocalandro, Evita Pueblo, Sanatorio Antartida, Hospital Central de San Isidro, Clinica Olivos in the state of Buenos Aires with 38 regional and town hospitals acting as referral centers, and Hospital Militar Central, Sanatorio de Los Arcos, Hospital Universitario CEMIC, Sanatorio Sagrado Corazon, Sanatorio Finochietto, Sanatorio Anchorena, Centro Gallego, and in the city of Buenos Aires in Argentina.

Study population. Subjects >= 75 years of age irrespective of presenting comorbidities or between 65-74 years of age with at least one comorbidity (hypertension, diabetes, obesity, chronic renal failure, and COPD) who experience the following signs and symptoms for less than 48 hours at the time of screening for SARS CoV2 by RT-PCR: (a) a temperature >=37.5°C and/or unexplained sweating and/or chills and (b) at least one of the following: dry cough, dyspnea, fatigue, myalgia, anorexia, sore throat, loss of taste and/or smell, rhinorrhea. Subjects consenting to screening will be tested by reverse-transcriptase-polymerase-chain-reaction (RT-PCR) for SARS-CoV-2 in a nasopharyngeal and an oropharyngeal swab and invited to participate when RNA for the virus is detected.

Intervention. Eligible, consenting patients will be randomized using an electronic system to receive 250 ml of convalescent plasma with an IgG titer against SARS-CoV2 spike (S) protein >1:1,000 (COVIDAR IgG, Insituto Leloir, Argentina) or placebo (normal saline 0.9%) administered in a 1:1 ratio. Both treatment and placebo will be concealed using dark bags and tape to cover the infusion line. Treatment will be administered <72 hours from initiation of symptoms. Subjects will be monitored for 12 hours after treatment for adverse events.

Clinical and laboratory monitoring. All participating subjects will be admitted to the hospital upon enrollment. Twenty-four hours after completing the infusion, a sample of venous blood (5 ml) will be obtained from all participants to measure anti-S IgG SARS-CoV2 in serum (COVIDAR IgG, Leloir) and preserved at -20°C until completion of the study. Patient evolution will be assessed daily by study physicians during hospitalization until day 25 and/or at home until day 15, in the event of earlier discharge from the hospital. Study physicians will use predesigned questionnaires to collect clinical information. An Independent Data Safety Monitoring Board (DSMB) will supervise participating subjects during the study.

Endpoints. The primary endpoint of the trial is development of severe respiratory disease defined as a respiratory rate (RR)>30 and/or an O2 sat<93% when breathing room air determined using a predefined protocol. Three other clinical endpoints include (a) life threatening respiratory disease, defined as need for 100% oxygen supplementation and/or non-invasive or invasive ventilation and/or admission to intensive care; (b) critical systemic illness, defined as respiratory failure (PaO2/FiO2 ≤ 200 mm Hg) and/or shock and/or multiorganic distress syndrome; and (c) death.

Statistical analysis. The study is designed to have one interim analysis when the outcome results for 50% of the subjects is obtained. The minimally clinically important difference was set at a 40% relative reduction for an expected outcome rate of 50% in the control group reduced to 30% in the intervention group. A total sample size of 210 subjects (105 per trial arm) was estimated to have 80% power at a significance level (alpha) of 0.05 using a two-sided z-test with continuity correction.

Ethical considerations. The trial has been approved by the institutional review boards of participating institutions and the Central Ethics Committee of the state of Buenos Aires. The study will be conducted in accordance with the principles of the Declaration of Helsinki and the Good Clinical Practice guidelines of the International Conference on Harmonization. Written informed consent will be obtained from all patients for screening and enrollment.

ELIGIBILITY:
Inclusion Criteria:

- Age ≥ 75 or age 65-74 with at least 1 of the following comorbidities: arterial hypertension, diabetes, obesity, chronic obstructive pulmonary disease, heart disease, chronic kidney disease

* Last 48 hours: (A)Axillary temperature ≥ 37.5oC or febrile equivalent, combined with (a) dry cough and/or (b) breathing difficulty and/or (c) odinophagia and/or (d) anosmia/dysgeusia and/or (e) any of the following symptoms: fatigue, anorexia, myalgias or rhinorrhea.
* Confirmed diagnosis SARS-Cov2 by RT-PCR
* Give Informed consent

Exclusion Criteria:

* Severe respiratory disease
* Cardiac insufficiency,
* Chronic renal failure,
* Primary hypogammaglobulinemias,
* Myelodysplastic syndromes,
* Chronic linfoproliferative syndromes,
* Monoclonal gammapathies,
* Known hypersensitibility,
* Active cancer,
* HIV, HBV or HCV infection,
* Chronic administration of immunosuppressants,
* Body transplant history,
* Chronic liver disease, Chronic lung disease with oxygen requirement.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 165 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Development of severe respiratory disease defined as a respiratory rate (RR)>30 and/or an O2 sat<93% | From 12 hours post infusion to day 15 post infusion

SECONDARY OUTCOMES:
Life threatening respiratory disease | From 12 hours post infusion to day 25 post infusion
Critical systemic illness, defined as respiratory failure | From 12 hours post infusion to day 25 post infusion
Death | From 12 hours post infusion to day 25 post infusion
Combination of secondary outcomes #2 (Life threatening respiratory disease) and/or #3 (Critical systemic illness, defined as respiratory failure) and//or #4 (death) | From 12 hours post infusion to day 25 post infusion
Duration of oxygen support requirement in patients with covid-19 due to saturation in ambient air <93%. | From 12 hours post infusion to day 25 post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Fernando P Polack, MD, Study Director — Fundacion Infant
Locations (11):
- Argentina (11):
  - Hospital Militar Central, CABA, Buenos Aires
  - CEMIC, CABA, Buenos Aires
  - Centro de Investigacion Clinica OSECAC, CABA, Buenos Aires
  - Centro Gallego de Buenos Aires, CABA, Buenos Aires
  - Sanatorio Anchorena, CABA, Buenos Aires
  - Sanatorio de Los Arcos, CABA, Buenos Aires
  - Hospital "Simplemente Evita", González Catán, Buenos Aires
  - Hospital Especializado de Agudos y Crónicos "San Juan de Dios", La Plata, Buenos Aires
  - Clinica Olivos, Buenos Aires
  - Hospital Central de San Isidro, Buenos Aires
  - Hospital General de Agudos "Dr. Carlos Bocalandro", Buenos Aires

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Nurmi V, Knight C, Estcourt L, Hepojoki J, Lamikanra AA, Tsang HP, Roberts DJ, Polack FP, Simmonds P, Hedman K, Alvarez-Paggi D, Harvala H. The Relationship Between SARS-CoV-2 Neutralizing Antibody Titers and Avidity in Plasma Collected From Convalescent Nonvaccinated and Vaccinated Blood Donors. J Infect Dis. 2023 Aug 11;228(3):245-250. doi: 10.1093/infdis/jiad070. PMID 36967714
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Libster R, Perez Marc G, Wappner D, Coviello S, Bianchi A, Braem V, Esteban I, Caballero MT, Wood C, Berrueta M, Rondan A, Lescano G, Cruz P, Ritou Y, Fernandez Vina V, Alvarez Paggi D, Esperante S, Ferreti A, Ofman G, Ciganda A, Rodriguez R, Lantos J, Valentini R, Itcovici N, Hintze A, Oyarvide ML, Etchegaray C, Neira A, Name I, Alfonso J, Lopez Castelo R, Caruso G, Rapelius S, Alvez F, Etchenique F, Dimase F, Alvarez D, Aranda SS, Sanchez Yanotti C, De Luca J, Jares Baglivo S, Laudanno S, Nowogrodzki F, Larrea R, Silveyra M, Leberzstein G, Debonis A, Molinos J, Gonzalez M, Perez E, Kreplak N, Pastor Arguello S, Gibbons L, Althabe F, Bergel E, Polack FP; Fundacion INFANT-COVID-19 Group. Early High-Titer Plasma Therapy to Prevent Severe Covid-19 in Older Adults. N Engl J Med. 2021 Feb 18;384(7):610-618. doi: 10.1056/NEJMoa2033700. Epub 2021 Jan 6. PMID 33406353